CLINICAL TRIAL: NCT07191951
Title: Shanghai Clinical Cohort - Adrenal Disease
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine (Unknown); RenJi Hospital (Other); Shanghai Zhongshan Hospital (Other); Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Wang Weiqing, Director of the Department of Endocrinology, Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Other Study IDs: SHDC2025CCS022
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Adrenal Disease
MeSH Terms: conditions — Adrenal Gland Diseases | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenal cohort: Aged between 18 and 75 years; diagnosed with adrenal diseases, including primary aldosteronism, pheochromocytoma, Cushing's syndrome, congenital adrenal hyperplasia, adrenocortical carcinoma, etc.; in stable condition, capable of tolerating all examinations and follow-ups required by the study.
  Interventions: Other: Receive adrenal surgery, radiotherapy, and/or medication therapy based on diagnosis and subtype classification.

INTERVENTIONS:
Other: Receive adrenal surgery, radiotherapy, and/or medication therapy based on diagnosis and subtype classification. — Receive adrenal surgery, radiotherapy, and/or medication therapy based on diagnosis and subtype classification.

SUMMARY:
As a vital organ responsible for producing life-sustaining hormones, the adrenal gland is associated with a wide range of diseases. These diseases affect multiple systems throughout the body and carry a high rate of mortality and disability. Current diagnosis and treatment face several challenges: significant variability in hormone testing results, inaccurate localization via imaging techniques, unclear molecular characteristics of adrenal tumors, and difficulty in determining prognosis through pathology. Therefore, establishing a clinical research cohort for adrenal diseases is essential. Such a cohort will enable in-depth exploration of disease mechanisms, identification of disease subtypes, optimization of diagnostic criteria, evaluation of treatment efficacy, advancement of personalized medicine, and formulation of prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form
* Commitment to abide by the study procedures and cooperate with the implementation of the entire study process
* Patients diagnosed with adrenal diseases, including aldosteronism, Cushing's syndrome, pheochromocytoma, adrenocortical carcinoma, and congenital adrenal hyperplasia; regardless of whether they have received adrenal surgery, radiotherapy, and/or medication therapy
* Aged between 18 and 75 years

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from this study:
* Refuse to sign the informed consent form
* Patients without adrenal diseases
* Have specified diseases or conditions (physical or psychological, identified through physical examination) that warrant exclusion from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged between 18 and 75 years; diagnosed with adrenal diseases, including primary aldosteronism, pheochromocytoma, Cushing's syndrome, congenital adrenal hyperplasia, adrenocortical carcinoma, etc.; in stable condition, capable of tolerating all examinations and follow-ups required by the study. These patients receive adrenal surgery, radiotherapy, and/or medication therapy based on diagnosis and subtype classification.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Treatment Remission Rate | at least six months or more
Treatment Response Rate | at least six months or more

CONTACTS AND LOCATIONS:
Locations (1):
- Jiang yiran, Shanghai, China

IPD SHARING:
Plan to Share IPD: No